CLINICAL TRIAL: NCT01823211
Title: Heart Rate Variability, Microvolt T-wave Alternans and Cardiac Magnetic Resonance Imaging Analysis in Primary Preventive ImplantablE Cardioverter-defibrillator Recipients Profitability Trial - HAPPIER Trial
Brief Title: Profitability Trial in Primary Preventive Implantable Cardioverter-defibrillator Recipients
Acronym: HAPPIER
Status: Terminated | Type: Observational
Why Stopped: Problems with ensuring patient examinations defined in the protocol of the study
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital Olomouc (Other); Brno University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KVO-2; Plasek680-2 (Registry Identifier: www.happiertrial.org)
Record Dates: First submitted 2013-03-19; First posted 2013-04-04 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Ischaemic Cardiomyopathy; Non-ischaemic Cardiomyopathy
Keywords: ICD (Implantable cardioverter-defibrillator); Heart rate variability; MTWA (Microvolt T-alternans); Magnetic resonance imaging (MRI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ischaemic cardiomyopathy: EP (Electrophysiology) study,magnetic resonance with LGE (Late gadolinium enhancement), ICD implantation
- non-ischaemic cardiomyopathy: EP study,magnetic resonance imaging with LGE, ICD implantation

SUMMARY:
The purpose of this study is further risk stratification of patients receiving implantable cardioverter-defibrillator in primary prevention of sudden cardiac death.

DETAILED DESCRIPTION:
Current criteria for risk stratification of patients in risk of sudden cardiac death are mainly based on left ventricular ejection fraction and NYHA class. This criteria are too robust, approximately 2/3 of ICD recipients do not profit from this treatment in the following 5 years, especially those with non-ischaemic cardiomyopathy. We plan to sub-stratify this group of patients with both ischaemic and non-ischaemic cardiomyopathy by: non-linear heart rate variability analysis, microvolt T-wave alternans, QRT-T angle and character and amount of left ventricular scarring assessed by magnetic resonance imaging. Pre-implantation values will be correlated with numbers and character of ICD therapy (both anti-tachycardial pacing and ICD discharge). The results may allow to decrease the number of patients, who do not profit from ICD treatment.

ELIGIBILITY:
Inclusion Criteria:

* LVD (left ventricular dysfunction) d/t MI (Myocardial infarction), LVEF 30% or less, NYHA (New York Heart association class) II, III
* LVD d/t MI, LVEF 30% to 35%, NYHA II, III
* LVD d/t MI, LVEF 30% to 40%, NSVT, positive EP study
* LVD d/t MI, LVEF 30% or less, NYHA I
* NICM (non-ischaemic cardiomyopathy), LVEF 30% or less, NYHA II, III
* NICM, LVEF 30% to 35%, NYHA II, III
* NICM, LVEF 30% or less, NYHA I
* signed informed consent

Exclusion Criteria:

* metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain, cannot have an MRI scan since the magnetic field may dislodge the metal
* severe claustrophobia may not be able to tolerate an MRI scan
* heart rhythm device in place before enrollment
* atrial fibrillation in time of enrollment
* ICD implantation indicated from secondary prevention of SCD (sudden cardiac death)
* NYHA or CCS class IV
* PCI or CABG in last 3 months
* CMP/TIA in last 3 months
* syncope of unknown etiology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart-failure clinic,primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
ventricular tachyarrhytmia | 36 months
  ventricular tachycardia equal or > 250/min,ventricular fibrillation, arrhythmic storm

SECONDARY OUTCOMES:
sudden cardiac death | 36-months
  death in 24-hours after symptom onset

OTHER OUTCOMES:
all-cause mortality | 36-months
  mortality from both cardiovascular and non-cardiovascular cause
Cardiovascular mortality | 36-months
  death from strictly cardiovascular cause

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Plasek, MD, PhD, Study Director — Department of Cardiology,University hospital Ostrava; Milos Taborsky, MD, PhD, FESC, Study Chair — Department of Cardiology,University Hospital Olomouc; Lubos Krivan, MD, PhD, Principal Investigator — Department of Cardiology,University Hospital Brno-Bohunice; Ondrej Moravec, MD, Principal Investigator — Department of Cardiology,University Hospital Olomouc
Locations (3):
- Czechia (3):
  - Brno University Hospital, Brno
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava

REFERENCES:
- [Background] Seely AJ, Macklem PT. Complex systems and the technology of variability analysis. Crit Care. 2004 Dec;8(6):R367-84. doi: 10.1186/cc2948. Epub 2004 Sep 22. PMID 15566580
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 guidelines for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Develop guidelines for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death) developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Europace. 2006 Sep;8(9):746-837. doi: 10.1093/europace/eul108. Epub 2006 Aug 25. No abstract available. PMID 16935866